## **Consent form template**

The consent form template below will be suitable for many studies but may need alterations to be commensurate with your study and must be used in conjunction with the guidance given in *Information Sheets & Consent Forms. Guidance for Researchers and Reviewers* 

For some studies a fuller, itemised or hierarchical consent form may be needed to cover important issues, especially if additional elements are optional for the participant. These may include:

- additional invasive tests or samples required for study purposes only;
- consent to use of audio/video-taping, with possible use of verbatim quotation or use of photographs;
- transfer of data/samples to countries with less data protection;
- agreement to receive individual feedback from testing.

| Centre Number: | | | | | |
|---|---|---|---|---|---|
| Stu | udy Number: | | | | |
| Pa | tient Identification Number fo | or this trial: | | | |
| | CONSE | NT FORM FOR PRE | GNANT \ | /OLUNTEERS | |
| Tit | le of Project: | | | | |
| | Serum blood clotting cha | anges during blood s | ampling v | ia non-luer one way filter va | alve |
| | intravenous need | le: Implications on th | e epidura | l blood patch procedure | |
| Name of Researcher: Dr Paul Sharpe Please | | | | Please initial | all boxes |
| 1. | I confirm that I have read at [2]) for the above study. I have had the | nave had the opportuni | ty to consi | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | |
| 4. | I agree for the research team to take blood samples from me with needles for the purposes of this study | | | | |
| 5. | I agree to my GP being informed if any abnormalities are found. | | | | |
| 6. | 6. I agree to take part in the above study. | | | | |
| | me of Participant | Date | | Signature | |
| Name of Person | | | | Signature | |

Consent form date of issue: [30/7/16] Consent form version number: [2]

taking consent.